CLINICAL TRIAL: NCT03486028
Title: Comparative Study Effectiveness of Clinical Decision-Making Processes Required by Public Health Systems Study
Brief Title: Patient Centered Assessment and Substance Use Disorder Treatment Study (PCAST)
Acronym: PCAST
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: University of California Integrated Substance Abuse Programs (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 0216289
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Substance Use Disorders
Keywords: Patient-Centered Outcomes Research Institute (PCORI); American Society of Addiction Medicine (ASAM); substance use; addiction; treatment; RTI International; UCLA
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASAM Counties/non-computerized: Pre- and 1115-waived counties that are implementing the ASAM. Intervention is adherence to ASAM protocols.
  Interventions: Other: Adherence to ASAM protocols
- ASAM Counties/computerized: Counties using a computerized system to assist in intervention determination according to ASAM protocols. Intervention is adherence to ASAM protocols.
  Interventions: Other: Adherence to ASAM protocols
- Non-ASAM Counties: Pre- and non-waived "control" counties that are not implementing the ASAM. Intervention is non-adherence to ASAM protocols.
  Interventions: Other: Non-adherence to ASAM protocols

INTERVENTIONS:
Other: Adherence to ASAM protocols — ASAM Counties. These counties are requiring their providers to use ASAM criteria to assess patients and to determine level of care. These counties also use ASAM to determine the ongoing need for high-intensity services, such as residential, and approve those services for Medicaid payment.
  Groups: ASAM Counties/computerized; ASAM Counties/non-computerized
Other: Non-adherence to ASAM protocols — These counties are not implementing the ASAM criteria to assess patients and determine the level of care.
  Groups: Non-ASAM Counties

SUMMARY:
California counties are in the process of implementing a Centers for Medicare and Medicaid Services Medicaid 1115 Substance Use Disorder (SUD) demonstration. The demonstration requires that patients be assigned to addiction treatment settings and levels of care systematically, using comprehensive biopsychosocial assessments and guided by the American Society of Addiction Medicine (ASAM) patient placement criteria.

RTI International, a nonprofit research institute, and University of California Los Angeles (UCLA) Integrated Substance Abuse Programs have been awarded a contract from the Patient Centered Outcomes Research Institute (PCORI) to study the effects of the ASAM implementation in California. The California 1115 SUD demonstration provides a unique opportunity to learn about the benefits and challenges resulting from system-wide implementation of ASAM criteria.

The study will involve surveying patients in counties that are using the ASAM criteria and in counties that have not yet adopted the ASAM criteria. Medicaid patients receiving addiction treatment will be offered the opportunity participate in the study and to be surveyed about their experiences in treatment. The study will also analyze data from the California Outcomes Management System (CalOMS) and conduct interviews with providers, patients, and policymakers in the state. The results of the study will help inform California's efforts to continually improve its addiction treatment systems to better meet the needs of it communities. This study will also produce important and useful information to patients seeking treatment for addiction, and their providers, SUD system administrators, and payers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 19 or older
* Receiving treatment for addiction in specialty addiction treatment programs licensed in California who are Medicaid beneficiaries.

Exclusion Criteria:

* Less than 19 years old
* Not receiving treatment for addiction in specialty addiction treatment programs licensed in California
* Not Medicaid beneficiaries

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals age 19 or older receiving treatment for addiction in specialty addiction treatment programs licensed in California who are Medicaid beneficiaries.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Treatment Retention | Up to one year
  Retention in treatment for at least 14 days is a validated outcome measure and has been shown to be predictive of reduced substance use, 2-year mortality, criminal justice involvement, and detox episodes. Retention in treatment can be measured with the CalOMS data.
Substance Use Reduction | Up to one year
  Abstinence and reduction in substance use is necessary for patients to achieve recovery and improved psychosocial functioning. We will measure this patient reported outcome (PRO) using the patient survey and CalOMS data. Through the patient survey, we will ask about use of any alcohol in the past 30 days, use of any drugs in the last 30 days, and the number of heavy drinking days in the last 30 days. These data will be collected from patients 3 months from treatment-episode initiation. Substance use is also collected from all patients treated in public SUD clinics in California at the beginning and end of each treatment episode and is recorded into the CalOMS data.

SECONDARY OUTCOMES:
Treatment setting used at treatment initiation | Up to one year
  Use of the ASAM criteria is anticipated to improve treatment outcomes (i.e., treatment retention and substance use) by increasing the use of more appropriate treatment settings for each patient, such as shifting the number of patients using residential, intensive outpatient, and opioid treatment programs. The treatment setting of each patient is tracked in the CalOMS data. Specifically, use of the following types of care is captured: (1) outpatient treatment, (2) intensive outpatient treatment, (3) outpatient detoxification, (4) residential detoxification (non-hospital), (5) residential detoxification (hospital), (6) residential treatment (30 days or less), and (7) residential treatment (30 days or more). Using the CalOMS data, we will test whether the distribution of the treatment setting used at treatment initiation changes after ASAM implementation.
Treatment option communication | Up to one year
  It is expected that ASAM implementation will improve communication from providers to patients about treatment options. We will assess this outcome through the patient survey.

CONTACTS AND LOCATIONS:
Overall Officials: Tami Mark, PhD, MBA, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No